CLINICAL TRIAL: NCT04236492
Title: Study Protocol for a Prospective Observational Study to Evaluate the Clinical and Imaging Results of the Fresh Osteochondral Allograft Transplantation for Osteochondral Knee Lesions
Brief Title: Study Protocol to Evaluate Clinical and Imaging Results of Knee Fresh Osteochondral Allografts
Status: Recruiting | Type: Observational
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Collaborators: Banc de Sang i Teixits (Other)
Responsible Party: Sponsor
Other Study IDs: IIBSP-ALO-2018-21
Record Dates: First submitted 2018-07-31; First posted 2020-01-22 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Osteochondral Defect
Keywords: fresh osteochondral allografts; integration; osteochondral defect; knee; chondral lesion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Fresh osteochondral allografting: Transplantation of a fresh osteochondral allograft in the knee
  Interventions: Procedure: Fresh osteochondral allografting

INTERVENTIONS:
Procedure: Fresh osteochondral allografting — Transplantation of a fresh osteochondral allograft in the knee

SUMMARY:
The main objective of this study is to assess the clinical and radiological results after carrying out a transplant of fresh osteochondral allograft in the knee.

DETAILED DESCRIPTION:
Fresh osteochondral allograft transplantation allows treatment of large osteochondral lesions of the knee in young patients. Real-world, patient-centered data on clinical and imaging results after fresh osteochondral allograft transplantation are needed.

This study is a prospective, observational, unicenter, patient-centered outcomes research study. Patients undergoing cartilage repair with fresh osteochondral allograft transplantation for osteochondral knee lesions are eligible to participate.

Clinical results are evaluated from baseline to 3 months, 6 months, 9 months, 12 months and 15 months postoperatively. At each time point, participants respond to several patient-reported outcome instruments to measure clinical results (IKDC, Kujala, Womet and Tegner) and patient satisfaction is captured.

Imaging results are evaluated with MRI (9 months and 15 months postoperatively) using the OCAMRISS evaluating cartilage features, bone features and ancillary features; and with CT (1 day, 3 months, 6 months and 12 months postoperatively) evaluating subchondral bone and osseous integration.

Variations will be explored using additional or alternative covariates such as concomitant surgery procedures, osteochondral allograft morphology, age, sex at birth, IMC, living situation and employment status.

ELIGIBILITY:
Inclusion Criteria:

Patients undergoing cartilage repair with fresh osteochondral allograft transplantation for large focal full-thickness chondral and osteochondral defects (>2 cm2) on the tibial plateau, femoral condyles, trochlea and/or patella Bipolar lesions are included.

Exclusion Criteria:

* BMI> 30 kg / m2
* Systemic inflammatory diseases
* Inflammatory arthritis
* Advanced osteoarthritis
* Tricompartmental degenerative process
* Active infection
* Patients who are unable to provide written informed consent.

Ages: 15 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Specialized care
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2018-06-06 (Actual); Primary Completion 2026-03-10 (Estimated); Study Completion 2026-11-10 (Estimated)

PRIMARY OUTCOMES:
International Knee Documentation Committee (IKDC) Score | 15 months
  The IKDC is a patient-completed tool, which contains three domains divided on 18 (7 items for symptoms, 1 item for sport participation, 9 items for daily activities, and 1 item for current knee function). Scores range from 0 points (lowest level of function or highest level of symptoms) to 100 points (highest level of function and lowest level of symptoms).
Kujala Score | 15 months
  The Kujala score is a 13-item questionnaire for the patient-reported assessment of anterior knee pain. The Kujala score asks about the ability to do several activities (squatting, stair climbing, running) and also the presence of symptoms/disabilities as noticed by the patient (limping, thigh atrophy, swelling, etc.). The items are summed up to give a total score ranging from 0 to 100, with high scores indicating good outcome.
Western Ontario Meniscal Evaluation Tool (WOMET) | 15 months
  WOMET is a disease-specific health-related quality of life questionnaire to measure physical symptoms, sports/reaction/work/lifestyle, and emotions of patients with meniscal pathology. It has 16 items representing the domains of physical symptoms (nine items), sports/recreation/work/lifestyle (four items), and emotions (three items). Lower scores indicate better outcome.
Tegner Activity Scale | 15 months
  Tegner activity level scale is a scale that aims to provide a standardized method of grading work and sporting activities. The patient selects the level of participation that best describes their current level of activity. A score of 0 represents "sick leave or disability pension because of knee problems," whereas a score of 10 corresponds to participation in national and international elite competitive sports. Activity levels 6-10 can only be achieved if the person participates in recreational or competitive sport.
Patient satisfaction | 15 months
  Patient satisfaction was captured using a 4-item categorical scale, with responses including extremely satisfied (4), satisfied (3), somewhat dissatisfied (2) and dissatisfied (1).
OCAMRISS | 15 months
  MRI will be performed at 9 and 15 months postoperatively. All MRI scans will be assessed by a musculoskeletal radiologist blinded to the patient's medical history and treatment using the OCAMRISS.
Bone integration | 15 months
  CT will be performed at 1 day postoperatively and at 3 months postoperatively, 6 months postoperatively and 12 months postoperatively. All CT scans will be assessed by a musculoskeletal radiologist blinded to the patient's medical history and treatment evaluating the subchondral bone and osseous integration. Collimation will be done in all CT to increase image quality and reduce the patient's overall radiation exposure.

SECONDARY OUTCOMES:
Age | 15 months
  Years
Sex at birth | baseline
  Man or female
IMC | baseline
  kg/m^2
Concomitant procedures | At the surgery
  Concomitant procedures (osteotomy, ligamentous repair/reconstruction, meniscal allograft transplantation) are recorded at the time of surgery.
Osteochondral allograft type | At the surgery
  Patellar, femoral or tibial

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Gelber, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Catalonia, Spain

REFERENCES:
- [Background] Flanigan DC, Harris JD, Trinh TQ, Siston RA, Brophy RH. Prevalence of chondral defects in athletes' knees: a systematic review. Med Sci Sports Exerc. 2010 Oct;42(10):1795-801. doi: 10.1249/MSS.0b013e3181d9eea0. PMID 20216470
- [Background] Mankin HJ. The response of articular cartilage to mechanical injury. J Bone Joint Surg Am. 1982 Mar;64(3):460-6. No abstract available. PMID 6174527
- [Background] Sherman SL, Garrity J, Bauer K, Cook J, Stannard J, Bugbee W. Fresh osteochondral allograft transplantation for the knee: current concepts. J Am Acad Orthop Surg. 2014 Feb;22(2):121-33. doi: 10.5435/JAAOS-22-02-121. PMID 24486758
- [Background] Widuchowski W, Widuchowski J, Trzaska T. Articular cartilage defects: study of 25,124 knee arthroscopies. Knee. 2007 Jun;14(3):177-82. doi: 10.1016/j.knee.2007.02.001. Epub 2007 Apr 10. PMID 17428666
- [Background] Bugbee WD, Convery FR. Osteochondral allograft transplantation. Clin Sports Med. 1999 Jan;18(1):67-75. doi: 10.1016/s0278-5919(05)70130-7. PMID 10028117
- [Background] Oakeshott RD, Farine I, Pritzker KP, Langer F, Gross AE. A clinical and histologic analysis of failed fresh osteochondral allografts. Clin Orthop Relat Res. 1988 Aug;(233):283-94. PMID 3042234
- [Background] Czitrom AA, Keating S, Gross AE. The viability of articular cartilage in fresh osteochondral allografts after clinical transplantation. J Bone Joint Surg Am. 1990 Apr;72(4):574-81. PMID 2324145
- [Background] Maury AC, Safir O, Heras FL, Pritzker KP, Gross AE. Twenty-five-year chondrocyte viability in fresh osteochondral allograft. A case report. J Bone Joint Surg Am. 2007 Jan;89(1):159-65. doi: 10.2106/JBJS.E.00815. No abstract available. PMID 17200323
- [Background] Sirlin CB, Brossmann J, Boutin RD, Pathria MN, Convery FR, Bugbee W, Deutsch R, Lebeck LK, Resnick D. Shell osteochondral allografts of the knee: comparison of mr imaging findings and immunologic responses. Radiology. 2001 Apr;219(1):35-43. doi: 10.1148/radiology.219.1.r01ap0435. PMID 11274532
- [Background] Gross AE, Kim W, Las Heras F, Backstein D, Safir O, Pritzker KP. Fresh osteochondral allografts for posttraumatic knee defects: long-term followup. Clin Orthop Relat Res. 2008 Aug;466(8):1863-70. doi: 10.1007/s11999-008-0282-8. Epub 2008 May 9. PMID 18465182
- [Background] Torga Spak R, Teitge RA. Fresh osteochondral allografts for patellofemoral arthritis: long-term followup. Clin Orthop Relat Res. 2006 Mar;444:193-200. doi: 10.1097/01.blo.0000201152.98830.ed. PMID 16523140
- [Background] Chu CR, Convery FR, Akeson WH, Meyers M, Amiel D. Articular cartilage transplantation. Clinical results in the knee. Clin Orthop Relat Res. 1999 Mar;(360):159-68. PMID 10101321
- [Background] Jamali AA, Emmerson BC, Chung C, Convery FR, Bugbee WD. Fresh osteochondral allografts: results in the patellofemoral joint. Clin Orthop Relat Res. 2005 Aug;(437):176-85. PMID 16056047
- [Background] Locht RC, Gross AE, Langer F. Late osteochondral allograft resurfacing for tibial plateau fractures. J Bone Joint Surg Am. 1984 Mar;66(3):328-35. PMID 6699046
- [Background] Shasha N, Krywulak S, Backstein D, Pressman A, Gross AE. Long-term follow-up of fresh tibial osteochondral allografts for failed tibial plateau fractures. J Bone Joint Surg Am. 2003;85-A Suppl 2:33-9. doi: 10.2106/00004623-200300002-00005. PMID 12721343
- [Background] Zou S, Dodd RY, Stramer SL, Strong DM; Tissue Safety Study Group. Probability of viremia with HBV, HCV, HIV, and HTLV among tissue donors in the United States. N Engl J Med. 2004 Aug 19;351(8):751-9. doi: 10.1056/NEJMoa032510. PMID 15317888